CLINICAL TRIAL: NCT03234829
Title: Determination of The Combined Mesio-Distal Widths of The Permanent Mandibular Incisors and That of The Maxillary and Mandibular Canines and Premolars in a Group of Egyptian Children in Rural Areas of Sohag Governorate: A Cross Sectional Study
Brief Title: Determination of Teeth Size in a Group of Egyptian Children. A Cross Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Atef, oral and dental medicine, principle investigator, Cairo University
Other Study IDs: MAtef
Record Dates: First submitted 2017-07-27; First posted 2017-07-31 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Teeth Size in a Group of Egyptian Children
Keywords: arch lengths, space analysis, arch prediction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Determination of The Combined Mesio-Distal Widths of The Permanent Mandibular Incisors and That of The Maxillary and Mandibular Canines and Premolars in a Group of Egyptian Children in Rural Areas of Sohag Governorate: A Cross Sectional Study

DETAILED DESCRIPTION:
Study Settings:

* Students will be randomly selected from preparatory schools in rural areas of Sohag governorate, seated in the school lap or an empty classroom.
* Clinical examination will be made in the daylight using disposable diagnostic sets (mirror, and explorer). No diagnostic radiographs will be taken.
* Operator: Master degree's student in Pediatric Dentistry and Dental Public Health.
* Full mouth alginate impression will be taken and study models will be poured within one hour with hard dental stone for each subject.
* Mesio-distal widths of both maxillary and mandibular permanent incisors, canines, first and second premolars will be measured from the study models using digital caliper according to the method described by(Moorrees & Reed, 1964) by measuring the greatest distance between the contact points on the proximal surfaces holding the caliper parallel to both occlusal and vestibular surfaces of the tooth.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are apparently medically free from any systemic disease.
2. Patients aged between 12-15 years.
3. Full set of fully erupted permanent dentition from left 1st permanent molar to right 1st permanent molar.
4. No apparent orthodontics problem.

Exclusion Criteria:

1. Patients with craniofacial developmental abnormality.
2. Any sensitivity or adverse reactions to any of used materials.
3. Patients who refused to participate in the study.
4. Teeth with severe malalignment or rotation.
5. Teeth with any inaccuracy caused by impression taking, pouring impressions with dental stone or any damage or breakage while the dental casts had been stored.
6. Teethwith notable wear, proximal decay, restorations, enamel hypoplasia or crown fracture.
7. Teeth with developmental anomalies such as microdont teeth, teeth with extra cusps or big talon cusps, or peg or conical shaped teeth.
8. Supernumerary or supplemental teeth (if present)

Ages: 12 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Students will be randomly selected using simple random sampling from preparatory schools in rural areas of Sohag governorate.
Sampling Method: Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The combined mesio-distal widths of the permanent mandibular incisors, the maxillary canines, mandibular canines and premolars. | one weak
  using Digital Caliper the data will be recorded in Millimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Eman S Elmasry, ass. prof, Study Director — Cairo University
Locations (1):
- Oral and Dental Medicine Faculity, Cairo, Egypt

REFERENCES:
- [Background] Shaweesh AI. Mesiodistal and faciolingual diameters of the permanent teeth in a Jordanian population. Arch Oral Biol. 2017 Jan;73:253-258. doi: 10.1016/j.archoralbio.2016.10.026. Epub 2016 Oct 26. PMID 27810383